CLINICAL TRIAL: NCT05689697
Title: Efficacy of Physiological Ketosis Induced by Liquid Technology Formula PanTrek in Asthenia and\or Decreased Tolerance to Physical and\or Mental Exertion (Double-blind, Placebo-controlled Study)
Brief Title: Induced Physiological Ketosis in Asthenia and\or Decreased Tolerance to Physical and\or Mental Exertion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ketonic Pharm LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KetonicPharm
Record Dates: First submitted 2022-12-23; First posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-12

CONDITIONS: Patient Activation
Keywords: Physiological Ketosis; PanTrek; Asthenia; Physical functioning; Mental functioning; beta-oxibutiric acid
MeSH Terms: conditions — Patient Participation; Asthenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: randomized asignment to placebo or IP group, double-blind design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): Patients will recieve matched by taste and color shot of 25 ml liquid in ampules
  Interventions: Dietary Supplement: PanTrek
- Active treatment group (Experimental): Patients will recieve shot of PanTrek 25 ml in anpules
  Interventions: Dietary Supplement: PanTrek

INTERVENTIONS:
Dietary Supplement: PanTrek — administration of exogenouse keton body

SUMMARY:
The purpose of this study is evaluating of efficacy of innovative dietary strategy -stimulation of physiological ketosis with Liquid Technology Formula PanTrek, in patients with asthenia and or decreased tolerance to physical and\or mental exertion. PanTrek is a liquid formula of potassium and magnesium salts of beta-oxibutiric acid, ginsenosides and rosmarinic acid.

DETAILED DESCRIPTION:
It will be double-blind, placebo-controlled study in 88 patients of both sex, aged from 18 to 65. Patients will be randomly assigned to one of two groups: placebo or IP group in 1:1 proportion. Study instruments: D-Fis, MoCA, TMT, VAS, assessment of blood keton concentration before and after first and last administration per os of 25 ml of placebo or PanTrek. PanTrek will be served in ampuls, 25 ml per ampule.

The duration of the study will be 15 days of treatment and 15 days of follow-up observation.

Patients will be assessed at screening/baseline, after 15 days and after 30 days.

The dose regimen: the shot of PanTrek, 25 ml, will be administered per os, twice per day, in the morning and in the evening, per se or deluted in 100 ml of water one hour before or after meal.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* diagnosis of astenia and/or decreased tolerance to physical and\or mental exertion
* ability of patients to understand assessment procedures

Exclusion Criteria:

* intollerance of components of PanTrek
* participation in other trials

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-01-09 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | 15 days
  Difference of changes of visual analog scale (VAS) indices between active treament and placebo groups. Minimum value - 0, maximum value - 100 scores. The higher score means the better condition. The major difference means better outcome.

SECONDARY OUTCOMES:
indused ketosis | 15 days
  increase of ketons level from baseline to the end of the active treatment period of the study

OTHER OUTCOMES:
Improvement in cognitive function | 15 days
  Difference in improvement in total scores of Montreal Cognitive Assessment (MoCA) between the treatment and placebo groups. Minimum value - 0, maximum value - 30 scores. The higher score means the better condition. The major difference means better outcome.
Improvement in visual attention and task switching. | 15 days
  Difference in improvement of total time of Trial Making Test (TMT) execution between the treatment and placebo groups. Normal value - 29 seconds for A part and 75 seconds for B part. The higher time means worse condition. Decrease of spended time means improvement or negative score, if the last result is substractes from the first result, means improvement.
Improvement in physical function | 15 days
  Difference in improvement in total scores of Daily Fatigue Investigation Scale (D-Fis) between the treatment and placebo groups. Minimum value - 0, maximum value - 32 scores. The higher score means the worse condition. The major difference means better outcome.
Safety profile in active and follow-up period | 30 days
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 on the first, 15th and 30th day.

CONTACTS AND LOCATIONS:
Overall Officials: Denis Burminskiy, MD, PhD, Study Director — Mental health research center
Locations (1):
- Laboratory of psychopharmacology Research center of mental health, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No